CLINICAL TRIAL: NCT05071261
Title: A Communication-Based Study Focused on Assessing and Improving Hepatitis C Screening Rates, As Well As Treatment Rates in Arizona as a Step Towards Disease Eradication
Brief Title: Screening, Treatment, and Eradication of Hep C
Status: Not yet recruiting | Type: Observational
Sponsor: Liver Institute PLLC (Other)
Responsible Party: Sponsor
Other Study IDs: LI-HEPC-AZ
Record Dates: First submitted 2021-09-16; First posted 2021-10-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Liver; Hepatitis C Virus; Screening; Disease Eradication
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hepatitis C Virus Screening — 1-2 Blood Screenings for Hepatitis C Virus

SUMMARY:
The aim of this study is to assess the HCV screening rate in Arizona by identification of potential HCV patients/subjects through different methods of communication - text message, email, social media, radio, newspaper ads, and flyers.

DETAILED DESCRIPTION:
The study will focus on various methods of communication to reach the population of Arizona from the most prevalent counties to lowest prevalence. The study is organized into phases focusing on the various communication methods beginning with direct communication through mass text messages and mass emails followed by indirect communication through social media (YouTube, Facebook), newspaper, radio, Alcoholics Anonymous meetings, Narcotics Anonymous meetings, and homeless shelters. Each phase will consist of four cycles of a monthly intervention period in which communication will be active and a two-month gap that will be used to assess effectiveness of the communication method. Subjects will receive information on HCV, contact information for the study coordinator at the Liver Institute PLLC to address questions or concerns, and a code that will allow them to receive a free HCV screening test at their local Sonora Quest Lab. This code can be used at the time of receipt or a few months later, whenever the subject is ready for testing. This timeline allows to enhance subject compliance. The results from Sonora Quest Lab will be transmitted to the study coordinator at the Liver Institute PLLC and depending on the subject's insurance status will link the subject to a treatment center. Ideally it will be their primary care physician but if the subject does not have one then it will be the closest treatment center. Alternatively, the Liver Institute PLLC is also equipped to provide telemedicine appointments to evaluate the subject and provide treatment depending on insurance status. Those that are uninsured will be provided with available options for treatment. All subjects will receive information on the disease to reduce transmission and encourage friends/family to get tested. This study will function on a version of the test-and-treat approach to help reduce the spread of HCV in the Arizona population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign the consent to screen and take part in the study.
* Subjects must be at least 15 years of age

Exclusion Criteria:

* Patients will only be enrolled once
* Patients who do not meet the inclusion criteria
* Patients with a current HCV diagnosis
* Patients who underwent a liver transplant

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All residents of Arizona
Sampling Method: Non-Probability Sample
Enrollment: 112136 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Screened | 5 years
  Number of subjects screened for HCV
Number of Subjects Treated | 5 years
  Number of subjects treated for HCV
Number of Subjects with a Positive Result for HCV | 5 years
  Number of subjects who received a positive test result for HCV

CONTACTS AND LOCATIONS:
Overall Officials: Huma Habib, MBA, Study Director — Director

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Background] 2016 Viral Hepatitis Epidemiologic Profile for Arizona (2016). Retrieved form https://www.azdhs.gov/documents/preparedness/epidemiology-disease-control/hepatitis/arizona-2016-viral-hepatitis-profile.pdf
- [Background] American Association for the Study of Liver Diseases (AASLD) and the Infectious Diseases Society of America (IDSA). (n.d.). Recommendations for testing, management, and treating hepatitis C. HCV testing and linkage to care. Retrieved from http://www.hcvguidelines.org
- [Background] Center for Disease Control and Prevention (CDC), (2016). Hepatitis C kills more Americans than any other infectious disease. Retrieved from https://www.cdc.gov/media/releases/2016/p0504- hepc-mortality.html
- [Background] Center for Disease Control and Prevention (CDC), (2018). Hepatitis C questions and answers for the public. Retrieved from https://www.cdc.gov/hepatitis/hcv/cfaq.htm#A1
- [Background] Chaffey, D. (2019) How do we compare? 2019 Email marketing statistics compilation. Retrieved from https://www.smartinsights.com/email-marketing/email-communications-strategy/statistics-sources-for-email-marketing/
- [Background] Denniston MM, Klevens RM, McQuillan GM, Jiles RB. Awareness of infection, knowledge of hepatitis C, and medical follow-up among individuals testing positive for hepatitis C: National Health and Nutrition Examination Survey 2001-2008. Hepatology. 2012 Jun;55(6):1652-61. doi: 10.1002/hep.25556. Epub 2012 Apr 10. PMID 22213025
- [Background] Hagan LM, Schinazi RF. Best strategies for global HCV eradication. Liver Int. 2013 Feb;33 Suppl 1(0 1):68-79. doi: 10.1111/liv.12063. PMID 23286849
- [Background] Homelessness. (n.d.). Retrieved from https://phoenixrescuemission.org/homelessness
- [Background] Holmberg SD, Spradling PR, Moorman AC, Denniston MM. Hepatitis C in the United States. N Engl J Med. 2013 May 16;368(20):1859-61. doi: 10.1056/NEJMp1302973. No abstract available. PMID 23675657
- [Background] Institute of Medicine (US) Committee on the Prevention and Control of Viral Hepatitis Infection; Colvin HM, Mitchell AE, editors. Hepatitis and Liver Cancer: A National Strategy for Prevention and Control of Hepatitis B and C. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK220039/ PMID 25032367
- [Background] Mappinghepc. (n.d.). Retrieved from https://mappinghepc.com/maps
- [Background] Palgrave-Jones, J. (2017). 5 Stats that prove 2017 is the year for SMS marketing. Retrieved from https://www.textlocal.com/blog/2017/06/16/5-stats-that-prove-2017-is-the-year-for-sms-marketing/
- [Background] Pinter M, Trauner M, Peck-Radosavljevic M, Sieghart W. Cancer and liver cirrhosis: implications on prognosis and management. ESMO Open. 2016 Mar 17;1(2):e000042. doi: 10.1136/esmoopen-2016-000042. eCollection 2016. PMID 27843598
- [Background] Snyder LB, Hamilton MA, Mitchell EW, Kiwanuka-Tondo J, Fleming-Milici F, Proctor D. A meta-analysis of the effect of mediated health communication campaigns on behavior change in the United States. J Health Commun. 2004;9 Suppl 1:71-96. doi: 10.1080/10810730490271548. PMID 14960405
- [Background] US Food and Drug Administration. (n.d.). FDA approves rapid test for antibodies to hepatitis C virus. News and Events. Retrieved from https://wayback.archive-it.org/7993/20170112215729/http:/www.fda.gov/NewsEvents/Newsroom/PressAnnouncement s/2010/ucm217318.htm
- [Background] Volk ML, Tocco R, Saini S, Lok AS. Public health impact of antiviral therapy for hepatitis C in the United States. Hepatology. 2009 Dec;50(6):1750-5. doi: 10.1002/hep.23220. PMID 19824079
- [Background] World Health Organization. (2018). Hepatitis C. Retrieved from https://www.who.int/news-room/fact-sheets/detail/hepatitis-c
- [Background] Yehia BR, Schranz AJ, Umscheid CA, Lo Re V 3rd. The treatment cascade for chronic hepatitis C virus infection in the United States: a systematic review and meta-analysis. PLoS One. 2014 Jul 2;9(7):e101554. doi: 10.1371/journal.pone.0101554. eCollection 2014. PMID 24988388

DOCUMENTS (2):
  • Study Protocol (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05071261/Prot_000.pdf
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05071261/ICF_001.pdf